CLINICAL TRIAL: NCT00844454
Title: Ethanol Ablation Using a Multi-pronged Needle and Radiofrequency Ablation of Early-stage Hepatocellular Carcinoma: a Randomized Clinical Trial
Brief Title: Multi-pronged Ethanol Ablation and Radiofrequency Ablation of Early-stage Hepatocellular Carcinoma
Acronym: QPEAvsRFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-de Lu, Department of Medical Ultrasound, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EARFArct; EARFArct2007
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; PEI; RF ablation; tumor ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QFEA (Experimental): multi-pronged ethanol ablation
  Interventions: Procedure: multi-pronged ethanol ablation
- RFA (Active Comparator): radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: multi-pronged ethanol ablation — Under ultrasound guidance, insert an applicator into the tumor percutaneously and then inject ethanol to destroy the whole tumor tissue.
  Arms: QFEA
Procedure: radiofrequency ablation — Under ultrasound guidance, insert an applicator into the tumor percutaneously and then deliver radiofrequency energy to destroy the whole tumor tissue.
  Arms: RFA

SUMMARY:
The purpose of this study is to compare the effectiveness of percutaneous ethanol ablation using a multi-pronged needle (QFEA) with that of percutaneous radiofrequency ablation (RFA) in the treatment of early-stage hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Patients with early-stage (single tumor no more than 5 cm or up to 3 tumors each no more than 3 cm in size) primary hepatocellular carcinoma will be randomized into two percutaneous ablation treatment arms, including radiofrequency ablation and multi-pronged ethanol ablation. The local treatment responses, complications,and long-term disease-free survivals and overall survivals are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Primary hepatocellular carcinoma, single tumor ≤5 cm or up to 3 tumors each ≤3 cm
* Ultrasound detectable tumor
* Liver function classified as Child-Pugh A or B
* Platelet count > 50,000/mm3, or prothrombin activity > 50%
* Not suitable for resection or patient refused surgery

Exclusion Criteria:

* Vascular invasion and extrahepatic spread
* Patients allergic to ethanol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Local treatment responses | 2 years

SECONDARY OUTCOMES:
Disease-free survivals and overall survivals | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mingde Lu, Prof., Principal Investigator — Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China